CLINICAL TRIAL: NCT06608264
Title: Effects of Stress Ball and Hand Holdig on Pain and Mobility Levels During Continuous Passive Motion In Patients With Total Knee Prosthesis: A Randomized Controlled Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, Rabia SARI, LECTURER, Necmettin Erbakan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 0517010149157
Record Dates: First submitted 2024-09-10; First posted 2024-09-23 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Pain and Mobility Levels of Patients Undergoing Total Knee Prosthesis During Continuous Passive Motion Exercise
Keywords: Pain, Knee Prosthesis, Patient Moving and Lifting, Nursing Care, Continuous Passive Motion Therapy.
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: Type of research:This study was planned as a randomized controlled experimental design to investigate the effects of stress ball and hand grip on pain and mobility levels during continuous passive movement in patients with TKA.
Who Masked: Outcomes Assessor
Masking Description: In order to prevent assignment bias in the study, blocks will be created by a statistician (in blocks of 6).The letters A, B, C representing the stress ball, hand grip and control arms will be determined by drawing lots.Since the researcher will be with the patient while performing the application, it will not be possible to blind the researcher during the application.However, the consultant will inform the researcher which patient is assigned to which arm once the patient meets the inclusion criteria and gives informed consent.The implementer will be blind to the appointment.The patient will be informed about which intervention (stress ball, hand holding, routine applications) will be performed after this stage. When entering the data into the SPSS database, the researcher will enter the data by coding the branches as A, B, C. Arms will not be reported to the statistician before reporting (blind technique)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control arm: (No Intervention): Patients who did not receive any intervention other than standard treatment and care during continuous passive motion exercise after total knee arthroplasty were defined as the control arm.
- stress ball arm (Experimental): Patients who underwent stress ball intervention during continuous passive motion exercise after total knee arthroplasty were defined as stress ball arms.
  Interventions: Other: stress ball intervention
- hand holding arm (Experimental): Patients who underwent hand-holding intervention during continuous passive range of motion exercise after total knee arthroplasty were defined as hand-holding arm.
  Interventions: Other: hand holding intervention

INTERVENTIONS:
Other: stress ball intervention — Stress ball intervention; A medium hard, round, high quality stress ball of the same brand will be given to the patient's actively used hand 1-2 minutes before starting the continuous passive movement exercise by the researcher.The patient will be asked to squeeze and relax the stress ball for a count of 5 during continuous passive movement.After squeezing the stress ball, the patient should count to 5 and then relax it.The patient will be asked to continue this process until the continuous passive movement exercise is completed.
  Arms: stress ball arm
Other: hand holding intervention — Hand holding intervention will be performed by the person the patient prefers. Before the continuous passive movement exercise, the person concerned will sit next to the patient's bed and warm their hands at a level that will not disturb the patient.1-2 minutes before the continuous passive motion exercise, the patient will hold the patient's hand with one hand, without using gloves, with moderate pressure, without rubbing or squeezing to an uncomfortable level.Hand holding intervention will continue until the continuous passive movement exercise is completed.
  Arms: hand holding arm

SUMMARY:
Pain after Total Knee Prosthesis (TKA) is an important problemWhen pain is not controlled, it can negatively affect the patients&#39; mobility level.This research; A randomized controlled experimental design was planned to examine the effects of stress ball and hand holding on pain and mobility levels in patients who underwent Continuous Passive Movement (CPM) after TOTAL knee prosthesis.The study was planned to be conducted between 15.07.2024 and 15.12.2025 on patients who who had total knee prosthesis surgery at the Aksaray University Training and Research Hospital Orthopedics and Traumatology Clinic.Since no study similar to our study design was found in the literature, the sample size of the study was calculated as 22 patients in each arm with Cohen* effect sizes for VAS, 3 arms, 2 repeated measurements, a medium effect size of 0.25 effect, 95% power and 5% type 1 error level.Considering that there may be data loss in the study, the sample size was increased by 20%, and a total of 78 patients, 26 in each arm.Assignment of patients to stress ball, hand holding and control arm using block randomization method,Determining by drawing lots which letters will represent the stress ball, hand holding and control arms as A, B, C,The blocks were planned to be created by a statistician."Stress ball intervention" to the stress ball arm during continuous passive movement exercise;&amp;amp;#34;Hand holding intervention&amp;amp;#34; will be made to the hand holding arm,"No intervention other than standard maintenance" will be made to the control arm.The implementation of the study will be carried out by the researcher R.S. and will be blinded to random assignment.On the 1st and 2nd days after total knee prosthesis, exercises are performed for 30 minutes with continuous passive movement.Considering this situation and the literature, the pain levels of the patients will be evaluated a total of 4 times on the 1st and 2nd days, before the CPM exercise, at the 5th minute, 15th minute and at the end of the exercise (30th minute); Mobility levels will be evaluated at this time, as the patient is mobilized within 1-2 hours after exercise.It was planned to collect the data with the "Patient Questionnaire Form, "Pain Assessment Form", "Patient Mobility Scale" and Observer Mobility Scale".Permission to use the scales was obtained via e-mail. Ethics committee and institution permissions were obtained to start the study.Data will be compared using Pearson chi-square, Fisher exact test, One-way ANOVA and repeated measures ANOVA, Kruskal Wallis test.It was planned to obtain informed consent from the patients before the study.The study is limited by the inclusion of patients with ASA I and II who underwent total knee prosthesis with a single physician and a single surgical technique at the Aksaray University Training and Research Hospital Orthopedics and Traumatology Clinic, regardless of whether they had chronic diseases.The study results can be used in planning the pain management of patients.It is thought that complications that may occur due to delayed mobilization and immobility can be prevented in patients whose pain is reduced.

DETAILED DESCRIPTION:
Type of research:This study was planned as a randomized controlled experimental design to investigate the effects of stress ball and hand holding on pain and mobility levels during continuous passive movement in patients with total knee prosthesis.

Research hypotheses:

H0 1: There is no difference in the pain levels of stress ball, hand holding and control arms during CPM in patients with total knee arthroplasty.

H1 1: There is a difference in the pain levels of stress ball, hand holding and control arms during CPM in patients with total knee prosthesis.

H0 2: There is no difference in the mobility levels of stress ball, hand holding and control arms during CPM in patients with total knee prosthesis.

H1 2: There is a difference in the mobility levels of stress ball, hand holding and control arms during CPM in patients with total knee prosthesis.

Universe of the research:The universe of the study will consist of patients who underwent total knee prosthesis in the Orthopedics and Traumatology Clinics of Aksaray University Training and Research Hospital.

Sample of the study: Since no study similar to our study design was found in the literature, the sample size of the study was calculated as 66 patients in total, 22 in each arm, with a medium effect size of 0.25 in 2 repeated measurements, 95% power and 5% type 1 error level, with 3 arms for Cohen* effect sizes for VAS. Considering that there may be data loss in the study, the sample size was increased by 20% in order not to decrease the statistical power, and a total of 78 patients, 26 in each arm (Suresh and Chandrashekara, 2012).

Collection of research data:

The Patient Questionnaire Form, which was developed by the researcher as a result of literature reviews (Dağcı, 2023; Khan et al., 2021; Ursavaş and Yaradılmış, 2021; Özbaş 2020; Yıldırım and Şendir, 2019; Mete and Avcı Işık, 2020), consists of seven questions to evaluate age, gender, marital status, education, employment, economic status and weight (Part I),It consists of two sections, namely, information on treatment and care (Section II), which consists of three questions on the presence of chronic diseases, ASA classification and patient examinations.

Pain Assessment Form was created to record the pain of patients before and during continuous passive exercise on the first and second day after total knee prosthesis by evaluating it with Visual Analog Scale: 4 stages.

Patient Mobility Scale: Scala was developed by Heye and his colleagues in 2002 and its validity and reliability study was conducted by Ayoğlu in 2011.The Patient Mobility Scale determines the level of pain and difficulty that patients will experience during any activity after surgery.After the surgical procedure, the pain and difficulty levels that patients develop while performing 4 activities such as turning from one side to the other in bed, sitting on the edge of the bed, standing up on the edge of the bed, and walking in the patient room are assessed with a 15 cm visual scale, which is verbally expressed by the patients.The degree of pain and difficulty of the patients is evaluated by measuring the distance between the mark they put on the scale and 0 with a calibrated ruler.Patients are asked 2 questions for each activity in the scale.Patients answer questions measuring the level and severity of pain perception using a five-point Likert-type scale [(1) no pain, (2) a little pain, (3) moderate pain, (4) a lot of pain, (5) the worst pain I could imagine], and the difficulty levels of the activities using a five-point Likert-type scale [(1) It was very easy, (2) It was easy, (3) It was a little difficult, (4) It was difficult, (5) It was very difficult].The lowest and highest scores that can be obtained from each item vary between 0-15, and the total scale score varies between 0-120.In the scale evaluation, an increase in the score indicates that the level of pain and difficulty during the implementation of the four activities increases.A decrease in the score indicates that the level of pain and difficulty in performing the four activities in patients decreases and the difficulty in moving decreases.

The Observer Mobility Scale, developed by Heye and colleagues in 2002, evaluates objective observations of movement during four activities in which patients perform postoperative activities, such as turning from one side to the other in bed, sitting at the edge of the bed, standing up at the edge of the bed, and walking in the patient room.Dependency/independence status is numbered from '1' to '5' A scale score of. '1' indicates that the person performs the relevant activity independently without verbal warning or physical assistance;The number '5' indicates that the patient is unable to perform the relevant activity despite verbal warning or physical assistance.Evaluation of the scale; the average score of the scale is obtained by summing the scores for the four activities that make up each item of the scale.Scores between 4 and 20 are obtained from the scale.As a result of the evaluation, an increase in the score indicates that the patients have a sufficient level of movement, and a decrease in the score indicates that the patients do not have a sufficient level of movement.

Research Data Collection:The research data were planned to be collected from patients who underwent total knee prosthesis in the Orthopedics and Traumatology Clinic between 20.09.2024 and 15.12.2025.Postoperative day 0: Continuous passive movement is not applied and the patient is not mobilized.On postoperative day I, patients will be evaluated according to inclusion and exclusion criteria by researcher RS.Patients who meet the inclusion criteria will be interviewed face to face to be informed about the research, and patients who volunteer to participate in the research will be asked to sign an Informed Consent Form.At this stage, it is not known by the researcher RS and the patient which group the patients will be included in. The "Patient Questionnaire Form" will be applied to all patients.After this stage, the arm to which the patient will be assigned (stress ball, hand holding and control arm) will be notified to the researcher by the consultant S.F. just before the intervention, according to the block randomization list created by the statistics expert.Just before the continuous passive exercise application, information will be given to the stress ball arm "regarding the stress ball application and data collection process"; and to the hand holding arm "regarding the hand holding application and data collection process".The control arm will only be given information about the "data collection process" and no intervention other than standard care will be made.

Stress ball intervention;A medium hard, round, high quality stress ball of the same brand will be given to the patient&amp;amp;#39;s actively used hand 1-2 minutes before starting the continuous passive movement exercise by the researcher.The patient will be asked to squeeze and loosen the stress ball for up to 5 counts during the continuous passive movement exercise.After squeezing the stress ball, the patient should count to 5 and then release it.The patient will be asked to continue this process until the continuous passive movement exercise is completed.

Hand holding intervention; It will be done by the person the patient prefers.Before the SPH exercise, the person concerned will sit next to the patient's bed and warm their hands to a level that will not disturb the patient.1-2 minutes before the continuous passive exercise, the patient will hold the patient's hand with one hand, without using gloves, with moderate pressure, without rubbing or squeezing to an uncomfortable level.Hand holding intervention will continue until the continuous passive movement exercise is completed.

The pain level of the patients during the continuous passive motion procedure will be evaluated with "VAS" in 4 stages, before the CPM exercise, at the 5th minute, at the 15th minute and at the end of the exercise (30th minute), with reference to the studies of Hsu et al. (2019) and Özgür and Rızalar (2021).The patient will mark the pain intensity on the 100 mm line 4 times on the "Pain Assessment Form". The mobility level of the patients will be evaluated with the "Patient Mobility Scale" and "Observer Mobility Scale" during the mobilization process after continuous passive motion exercise on the 1st and 2nd days after total knee prosthesis, in line with the literature review (Sütçü 2022, Danç 2019).

All patients are mobilized by the orthosis-prosthesis technician within 1-2 hours after continuous passive movement exercises.The Patient Mobility Scale and the Observer Mobility Scale will be applied during "Turning from One Side to the Other in Bed", "Sitting at the Edge of the Bed", "Standing at the Edge of the Bed" and "Walking in the Patient Room"For the Patient Mobility Scale, the patient is expected to mark on a 150 mm line the level of pain and difficulty he/she experiences after performing each of these four steps.The 4 activities that constitute the subgroup of patient mobility will be observed simultaneously by the researcher RS and the orthosis-prosthesis technician.The Observer Mobility Scale will be evaluated simultaneously by two observers at these stages and filled in according to common opinion.While filling out the Visual Analog Scale, Patient Mobility Scale and Observer Mobility ScaleThe markings made by the patient will be measured and recorded with the same ruler calibrated by the researcher after the procedure.Medical treatments for pain were standardized with the physician, taking into account the life of the drug (paracetamol) used.Application of treatment other than this standardized treatment before Continuous Passive Movement and mobilization has been added to the exclusion criteria. However, Patients who defined 4 or more pain levels after the procedure would be unethical to withhold analgesic treatment and Since it will not affect the Visual Analog Scale, Patient Mobility Scale and Observer Mobility Scale values used in the study, additional analgesic treatment can be applied.

Variables of the Study; Independent Variables:Hand holding application, stress ball application Dependent Variables:Pain levels, Patient Mobility Levels Ethical Aspects of the Research:Ethics Committee permission was obtained for the implementation of the research.Institutional permission was received from Aksaray Provincial Health Directorate to conduct the implementation phase of the research at Aksaray University Training and Research Hospital.Permission was obtained from Tuluha AYOĞLU via e-mail for the use of the Patient Mobility Scale and Observer Mobility Scale.Patients who will be included in the research will be informed that their research data will be used only for academic purposes.Preliminary information will be provided that all initiatives to be implemented are carried out in line with universal ethical principles.Informed Consent will be obtained verbally and in writing.

Limitations of the Study:The treatment and care process of the patients is shaped according to the routine practices of this hospital.Patients who underwent total knee prosthesis at the Orthopedics and Traumatology Clinic of Aksaray University Training and Research Hospital were included in the study.Limited to a single physician and a single surgical technique (paramedial arthrotomy). Since the possible chronic diseases of the patients cannot be predicted, whether they have chronic diseases or not is ignored.Taking the ASA assessment into account, ASA I and II patients were included in the study and those with III, IV and V were excluded, thus attempting to ensure similarity in the health status of the patients.

Statistical Evaluation of Data: Data will be evaluated in the statistical package program IBM SPSS Statistics 26.0 (IBM Corp., Armonk, New York, USA). Descriptive statistics will be given as number of units (n), percentage (%), mean±standard deviation, median, smallest value, largest value and percentile values.The normal distribution of data belonging to numerical variables will be evaluated with the Shapiro Wilk normality test.If the data show a normal distribution, Visual Anolaog Scale comparisons according to the measurement times of the arms will be made with Two-Way Analysis of Variance in Repeated Measurements from general linear models.Bonferroni correction will be applied to all pairwise comparisons.Observer and patient mobility scale scores obtained after 60 minutes of Continuous passive arm movement exercise will be compared using One-Way Analysis of Variance. If the Ho hypothesis is rejected in one-way analysis of variance, the Duncan test will be used as a multiple comparison test. If the data do not show a normal distribution, comparisons between arms are made using Kruskal-Wallis Analysis, Intra-arm comparisons will be made with Wilcoxon analysis. If a difference is found in the Kruskal-Wallis Analysis, the Dunn-Bonferroni test will be used as a multiple comparison test.Chi square analysis (Pearson chi square or Fisher exact test) will be used to compare the arms with categorical variables. p&amp;amp;amp;amp;amp;amp;lt;0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* After being informed about the study, written permission was obtained for voluntary participation
* Ages 18 and over
* In the preoperative evaluation, ASA scores were at levels I and II.
* Able to speak Turkish and communicate verbally

  * A combination of spinal anesthesia and adductor block was applied during the surgery.
  * first time and unilateral total knee prosthesis was performed
  * Total knee prosthesis surgery is performed by the same physician and the same surgical technique
* Patients who underwent continuous passive movement exercise after removing the hemovac drain on the first day after surgery were planned to be included in the study.

Exclusion Criteria:

* Alzheimer's, dementia-like conditions that prevent understanding
* Analgesic was administered outside of the analgesic treatment plan determined before continuous passive movement exercise.
* General anesthesia or a different anesthesia is applied during the surgery.
* Patients who stay in the recovery unit for more than 1 hour (more than the routine period) after surgery or who receive treatment and care in the intensive care unit (patients whose vital signs are unstable, who develop lung problems, who are bleeding, who require blood transfusion, who have severe pain)
* Describing pain outside the surgical area
* In the preoperative evaluation, it was planned that patients with ASA scores of III, IV and V would not be included in the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2024-09-25 (Estimated); Primary Completion 2025-06-25 (Estimated); Study Completion 2025-12-25 (Estimated)

PRIMARY OUTCOMES:
pain levels | Pain levels of the patients will be evaluated in 4 stages, including the 5th minute, 15th minute and 30th minute of the exercise, before the continuous passive movement exercise between 09:00 and 14:00 on the 1st and 2nd postoperative days.
  The pain level of the patients will be evaluated with Visual Analogue Scale (VAS)
Patient Mobility Levels checklist | Patient mobility levels will be assessed during the mobilization process (position change, sitting, standing up, walking) within 1-2 hours after continuous passive movement exercise,between 09.00-14.00 on the 1st and 2nd day after the surgery

CONTACTS AND LOCATIONS:
Overall Officials: Rabia SARI, LECTURER, Principal Investigator — AKSARAY UNIVERSITY/AKSARAY/TURKIYE; Saide FAYDALI, Associate Professor, Study Director — NECMETTIN ERBAKAN UNIVERSITY/KONYA/TURKIYE
Locations (1):
- Aksaray Training and Research Hospital [Aksaray Eğitim ve Araştırma Hastanesi], Aksaray, Aksaray/center, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No